CLINICAL TRIAL: NCT00300196
Title: ASP II (Ancrod Stroke Program) Study of Acute Viprinex™ for Emergency Stroke: A Randomized, Double-Blind, Placebo-Controlled Study of Ancrod (Viprinex™) in Subjects Beginning Treatment Within 6 Hours of the Onset of Acute Ischemic Stroke
Brief Title: ASP-II: Ancrod Stroke Program: Ancrod (Viprinex™) for the Treatment of Acute, Ischemic Stroke
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Neurobiological Technologies (Industry)
Responsible Party: Warren W. Wasiewski, M.D., Neurobiological Technologies, Inc. (no longer active)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTI-ASP-0503
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Stroke; Cerebral Ischemia; Brain Infarction
Keywords: Stroke; Fibrinogen; Reperfusion; Thrombolysis
MeSH Terms: conditions — Stroke; Brain Ischemia; Brain Infarction | interventions — Ancrod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous ancrod (Experimental): Intravenous ancrod infused at a rate of 0.167 IU/kg/hr (0.6 mL/kg/hr) for 2 or 3 hours depending on the pretreatment fibrinogen level.
  Interventions: Biological: Ancrod (Viprinex)
- Intravenous Placebo (Placebo Comparator): Intravenous placebo at a rate of 0.6 mL/kg/hr for 2 or 3 hours depending on the pretreatment fibrinogen level.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ancrod (Viprinex) — 0.167 IU/kg/hr IV for 2-3 hours
  Arms: Intravenous ancrod
Drug: Placebo — 0.6 mL/kg/hr
  Arms: Intravenous Placebo

SUMMARY:
The primary purpose of this study is to determine whether a brief intravenous infusion of ancrod started within 6 hours of stroke onset improves functional outcome at 3 months.

DETAILED DESCRIPTION:
With prior approval by the FDA, an interim analysis for futility was performed when 500 subjects had been entered into the two parallel trials, NCT00141001 and NCT00300196. The analyses were reviewed by the data safety monitoring board, which recommended that both studies be terminated because of futility. This was done at a point where 650 subjects had been entered into both studies, combined, but analyses were conducted only on the initial 500 subjects. Results of the abbreviated analysis will be found with study NCT00141001 since that study contributed most of the subjects to the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acute, ischemic stroke with first symptoms within 6 hours of beginning treatment
* Baseline NIHSS > 5

Exclusion Criteria:

* No intracranial, extravascular blood on CT
* Hypertension (systolic > 185; diastolic > 105)
* Baseline fibrinogen level < 100 mg/dL
* Thrombocytopenia (< 100,000 / mm3)
* Recent (< 3 days) or anticipated (< 5 days) use of a thrombolytic agent
* Recent (< 14 days) or anticipated surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Score - responder analysis | 90 days

SECONDARY OUTCOMES:
Barthel Index, NIHSS | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Warren Wasiewski, M.D., Study Director — Neurobiological Technologies
Locations (93):
- United States (39):
  - Enloe Medical Center, Chico, California
  - UCSF-Fresno, Fresno, California
  - Sherry Braheny MD - A Prof. Corporation, La Mesa, California
  - Mercy General Hospital, Sacramento, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Manatee Memorial Hospital, Bradenton, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Naples Community Hospital, Naples, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Joan Glancy Memorial Hospital, Decatur, Georgia
  - Joan Glancy Memorial Hospital, Duluth, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Dekalb Medical Center-Hillandale, Lithonia, Georgia
  - Candler Hospital, Savannah, Georgia
  - St. Joseph's Hospital, Savannah, Georgia
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Saint Luke's Hospital Mid America Brain and Stroke Institute, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - St. Louis University Hospital - Dept of Neurology, St Louis, Missouri
  - Nevada Neuroscience Institute at Sunrise, Las Vegas, Nevada
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Neuroscience Institute St Francis Medical Center, Trenton, New Jersey
  - Lutheran Medical Center, Brooklyn, New York
  - Five Towns Neuroscience Research, Lawrence, New York
  - Aultman Hospital, Canton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hahenmann University Hospital, Philadelphia, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Providence St. Peter Hospital, Olympia, Washington
  - CAMC Memorial Hospital, Charleston, West Virginia
- Australia (6):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Gold Coast Hospital, Southport, Queensland
  - Moash Medical Center Dept of Neurology, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Alfred Hospital Research - Melbourne, Prahan, Melbourne, Victoria
  - Concord Hospital Neuroscience Department, New South Wales
- Austria (2):
  - Medical University of Affairs, Graz
  - Neurologische Intensivstation, Linz
- Czechia (7):
  - University Hospital Hradec Kralove Neurological Department, Hradec Králové
  - PalackyUniversity Faculty of Medicine and Dentistry and University Hospital, Olomouc
  - Vitkovice Hospital Department of Neurology, Ostrava
  - Regional Hospital Pardubice, Pardubice
  - General University Hospital Clinic of Neurology-Stroke Center, Prague
  - Thomayer's Faculty Clinic of Neurology, Prague
  - University Hospital Motol Department of Neurology, Prague
- Israel (10):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center Dept of Neurology Ben-Gurion Univ of the Negev, Beersheba
  - Bnei-Zion Medical Center, Haifa
  - Rambam Medical Center Dept. of Neurology, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Ein-Karem Medical Center, Jerusalem
  - Western Galilee Hospital Neurology Dept, Nahariya
  - Rabin Medical Center Golda Campus (Hasharon), Petah Tikva
  - Tel-Aviv Medical Center, Tel Aviv
  - Chaim Sheba Medical Center Neurology Dept, Tel Litwinsky
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Cristchurch Hospitial, Christchurch
- Poland (5):
  - Samodzielny Publiczny Szpital Kliniczny nr1, Akademickie Centrum, Gdansk
  - Katedra i Klinika Neurologii, Wieku Podesziego, Katowice
  - Klinika Neurologii Akademii Medycznej w Lublinie, Lublin
  - Centrum Medycne HCP sp.zo.o Dept. Neurlogy, Poznan
  - Institute for Psychiatry and Neurology 2nd Neurology Dept., Warsaw
- Russia (12):
  - State Multiregional Clinical Diagnostical GU MKDZ, Kazan'
  - Central clinical Hospital of the President of the Russian Federation, Moscow
  - Burdenko Central Military Clinical Hospital of Ministry of Defense of Russia, Moscow
  - Municipal Institution of Health City Clinical Hospital No. 1, Novosibirsk
  - Hospital Baranov, Petrozavodsk
  - Railway Hospital at Rostov-Glavnity of OJSC "Russian Railways", Rostov-on-Don
  - Multiprofile City Clinic No. 2, Saint Petersburg
  - City Clinic Neurology N2 of Marinski Hospital, Saint Petersburg
  - State Medical University named after IP Pavlov Leo Tolstoj, Saint Petersburg
  - City Hospital Nr. 1 of Pirogov, Samara
  - Jaroslav Regional Clinical Hospital State Institution of Healthcare, Yaroslavl
  - City Clinical Hospital MU KGB Nr. 40, Yekaterinburg
- Slovakia (7):
  - Fakultna nemocnica s poliklinikou Bratislava, Bratislava
  - Vseobecna nemocnica s polokliniknikou Levoca a.s., Levoča
  - Martinska fakultna nemocnica, Martin
  - Fakultna nemocnica Nitra, Nitra
  - Nemocnica s poliklinikou Spisska, Nová Ves
  - Fakultna nemocnica s poliklinikou J.A. Reimana, Prestov
  - Fakultna nemocnica Trnava, Trnava
- Clinical Projects Research, Worcester, South Africa
- Switzerland (2):
  - Centre Hospitalier universitaire Vaudois, Dept. of Neurology, Lausanne
  - Universitatsspital Zurich, Zurich

REFERENCES:
- See also: Related Info — http://www.ntii.com